CLINICAL TRIAL: NCT07127523
Title: A Randomized, Triple-blind, Placebo Controlled, Parallel Virtual Clinical Trial to Investigate the Efficacy and Safety of GenLabs' Social Skin on Improving Acne Symptoms and Skin Repair Among Healthy Adults
Brief Title: A Clinical Trial to Investigate the Efficacy and Safety of GenLabs' Social Skin on Improving Acne Symptoms and Skin Repair Among Healthy Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GenCanna Acquisition Corp (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25GCCFT01
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-08

CONDITIONS: Acne
Keywords: GenLabs; Social Skin; Acne symptoms
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Skin (Experimental): The investigational product in this study contains ProRenew Complex CLRTM, which is a three-step skin regime targeting acne comprised of Lactococcus ferment lysate, derived from L. lactis, in addition to peppermint, willow bark, and lentil seed extracts. Apply the 3 study products in the morning and at night before bed. The participants will be required to maintain their application times throughout the study duration. Application of the study products covering the face and neck will occur in a step-wise fashion (Step 1, Step 2, Step 3) for 30 days.
  Interventions: Other: Social Skin
- Placebo (Placebo Comparator): This group receives a placebo containing non-medicinal ingredients in Social Skin, in a three-step skin regime. Apply the 3 study products in the morning and at night before bed. The participants will be required to maintain their application times throughout the study duration. Application of the study products covering the face and neck will occur in a step-wise fashion (Step 1, Step 2, Step 3) for 30 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Social Skin — This group receives a cleanser, serum, and cream.
  Arms: Social Skin
Other: Placebo — This group receives a cleanser, serum, and cream.
  Arms: Placebo

SUMMARY:
The goal of this interventional clinical trial is to investigate the efficacy and safety of GenLabs' Social Skin on improving acne symptoms and skin repair among healthy adults. The main question[s] it aims to answer is:

What is the difference in the change in acne symptoms as assessed by the Acne Quality of Life Questionnaire (ACNE-QoL) between GenLabs' Social Skin and placebo from baseline at Day 30.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 65 years of age inclusive
2. Females not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening

   Or,

   Individuals of child-bearing potential must self-report confirmation they are not pregnant, do not plan to become pregnant, and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
   * Abstinence
3. Experience acne on facial skin that is visible to the participant and is confirmed by the QI at screening and at baseline
4. Willingness to complete questionnaires and diaries associated with the study, to capture and upload photos, and to complete all virtual visits
5. Willingness to maintain the same skincare regimen throughout the study, including maintaining make-up routine without the addition of new make-up products
6. Agrees to maintain current lifestyle habits (diet, physical activity, medications, supplements, and sleep) as much as possible throughout the study
7. Provided voluntary, written, informed consent to participate in the study
8. Agrees to have de-identified photos of face available for marketing purposes
9. Self-reported healthy as determined by medical history with no unstable diagnosed medical conditions

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Self-reported allergy, sensitivity or intolerance to investigational product or placebo ingredients, including allergy to salicylic acid or any form of salicylates, preventing topical use
3. Individuals with significant facial hair that would impede the visualization of facial acne and may interfere with the use of the product, such as beards and long sideburns, as assessed by the QI
4. Self-reported psoriasis, dermatitis, vitiligo, or any other active dermatological condition other than acne affecting the face
5. Self-reported use of topical products on the face marked with claims relating to skin health, or those with claims relating to acne during the study, except for noncomedogenic moisturizers and sunscreen
6. Self-reported shaving, waxing, tweezing, or threading of the face or use of nose/facial strips within 3 days prior to each photo capture
7. Procedures such as microdermabrasion, peels, acne treatments, filler, botulinum toxin, red light therapy, pore suction therapy, or laser on the face within three months of baseline
8. Self-reported UVA or UVB exposure to the face in the past two weeks or expected during the study to avoid sunburn.
9. Current use of prescribed and/or over-the-counter (OTC) medications, supplements, and/or consumption of food/drinks that may impact the efficacy and/or safety of the investigational product (Sections 7.3.1 and 7.3.2)
10. Self-reported asthma
11. Self-reported presence of a peptic ulcer
12. Self-reported autoimmune disease or are immune compromised
13. Self-reported ongoing and unstable diseases/conditions in the past three months, including:

    1. Arthritis and joint diseases
    2. Gastrointestinal diseases
    3. Hypertension
    4. Type I or type II diabetes
    5. Cardiovascular disease
    6. Kidney diseases
    7. Liver diseases
    8. Thyroid condition
    9. Psychiatric conditions
14. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study
15. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
16. Alcohol intake average of >2 standard drinks per day
17. Alcohol or drug abuse within the last 12 months
18. Participation in other clinical research studies 30 days prior to screening
19. Individuals who are unable to give informed consent
20. Any other condition or lifestyle factor that may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The difference in the change in acne symptoms as assessed by the Acne Quality of Life Questionnaire (ACNE-QoL) between GenLabs' Social Skin and placebo | Day 0 to 30
  The difference in the change in acne symptoms as assessed by the Acne Quality of Life Questionnaire (ACNE-QoL) between GenLabs' Social Skin and placebo from baseline at Day 30. The Acne symptoms domain of the Acne-QoL is comprised of 5 questions which assess the physical symptoms experienced by facial acne sufferers. Questions include the number of bumps on the face, the extent of scabbing from the acne, and the level of worry associated with scarring from the acne.

SECONDARY OUTCOMES:
The difference in the change in acne symptoms as assessed by the Acne Quality of Life Questionnaire (ACNE-QoL) between GenLabs' Social Skin | Day 0 to 10
  The difference in the change in acne symptoms as assessed by the Acne Quality of Life Questionnaire (ACNE-QoL) between GenLabs' Social Skin and placebo from baseline at Day 10
The difference in the change in acne symptoms as assessed by the Acne Quality of Life Questionnaire (ACNE-QoL) between GenLabs' Social Skin | Day 0 to 20
  The difference in the change in acne symptoms as assessed by the Acne Quality of Life Questionnaire (ACNE-QoL) between GenLabs' Social Skin and placebo from baseline at Day 20.
The difference in change in acne symptoms as assessed by the Self-assessment of Clinical Acne-Related Scars (SCARS) between GenLabs' Social Skin and placebo | Day 0 to 10
  The difference in change in acne symptoms as assessed by the Self-assessment of Clinical Acne-Related Scars (SCARS) between GenLabs' Social Skin and placebo from baseline at Day 10. The SCARS has two parts, part 1 asks questions related to current active acne including zits, breakouts, pimpled, whiteheads, and blackheads, and questions related to atrophic scaring including indents or holes in the skin from previous active acne. Part 2 of the SCARS, assess acne scar appearance and severity with 5 questions such as how much of your face is covered by indents or holes with five potential answers: almost none of my face, a little of my face, some of my face, a lot of my face, and almost all of my face
The difference in change in acne symptoms as assessed by the Self-assessment of Clinical Acne-Related Scars (SCARS) between GenLabs' Social Skin and placebo | Day 0 to 20
  The difference in change in acne symptoms as assessed by the Self-assessment of Clinical Acne-Related Scars (SCARS) between GenLabs' Social Skin and placebo from baseline at Day 20. The SCARS has two parts, part 1 asks questions related to current active acne including zits, breakouts, pimpled, whiteheads, and blackheads, and questions related to atrophic scaring including indents or holes in the skin from previous active acne. Part 2 of the SCARS, assess acne scar appearance and severity with 5 questions such as how much of your face is covered by indents or holes with five potential answers: almost none of my face, a little of my face, some of my face, a lot of my face, and almost all of my face
The difference in change in acne symptoms as assessed by the Self-assessment of Clinical Acne-Related Scars (SCARS) between GenLabs' Social Skin and placebo | Day 0 to 30
  The difference in change in acne symptoms as assessed by the Self-assessment of Clinical Acne-Related Scars (SCARS) between GenLabs' Social Skin and placebo from baseline at Day 30. The SCARS has two parts, part 1 asks questions related to current active acne including zits, breakouts, pimpled, whiteheads, and blackheads, and questions related to atrophic scaring including indents or holes in the skin from previous active acne. Part 2 of the SCARS, assess acne scar appearance and severity with 5 questions such as how much of your face is covered by indents or holes with five potential answers: almost none of my face, a little of my face, some of my face, a lot of my face, and almost all of my face
The difference in change in self-perception, social impact, and emotional impact as measured by the ACNE-QoL between GenLabs' Social Skin and placebo | Day 0 to 10
  The difference in change in self-perception, social impact, and emotional impact as measured by the ACNE-QoL between GenLabs' Social Skin and placebo from baseline at Day 10
The difference in change in self-perception, social impact, and emotional impact as measured by the ACNE-QoL between GenLabs' Social Skin and placebo | Day 0 to 20
  The difference in change in self-perception, social impact, and emotional impact as measured by the ACNE-QoL between GenLabs' Social Skin and placebo from baseline at Day 10
The difference in change in self-perception, social impact, and emotional impact as measured by the ACNE-QoL between GenLabs' Social Skin and placebo | Day 0 to 30
  The difference in change in self-perception, social impact, and emotional impact as measured by the ACNE-QoL between GenLabs' Social Skin and placebo from baseline at Day 10
The difference in change in acne appearance as assessed by the participant and investigator using the Global Aesthetic Improvement Scale (GAIS) between GenLabs' Social Skin and placebo | Day 0 to 10
  The difference in change in acne appearance as assessed by the participant and investigator using the Global Aesthetic Improvement Scale (GAIS) between GenLabs' Social Skin and placebo from baseline at Day 10. The GAIS categorizes acne improvement according to a five-point scale (1 - Very much improved, 2 - Much improved, 3- Improved, 4- No change, 5- Worsened).
The difference in change in acne appearance as assessed by the participant and investigator using the Global Aesthetic Improvement Scale (GAIS) between GenLabs' Social Skin and placebo | Day 0 to 20
  The difference in change in acne appearance as assessed by the participant and investigator using the Global Aesthetic Improvement Scale (GAIS) between GenLabs' Social Skin and placebo from baseline at Day 20. The GAIS categorizes acne improvement according to a five-point scale (1 - Very much improved, 2 - Much improved, 3- Improved, 4- No change, 5- Worsened).
The difference in change in acne appearance as assessed by the participant and investigator using the Global Aesthetic Improvement Scale (GAIS) between GenLabs' Social Skin and placebo | Day 0 to 30
  The difference in change in acne appearance as assessed by the participant and investigator using the Global Aesthetic Improvement Scale (GAIS) between GenLabs' Social Skin and placebo from baseline at Day 30
The difference in change in acne scar appearance as assessed by the participant using the Vancouver Scar Scale (VSS) between GenLabs' Social Skin and placebo | Day 0 to 10
  The difference in change in acne scar appearance as assessed by the participant using the Vancouver Scar Scale (VSS) between GenLabs' Social Skin and placebo from baseline at Day 10. The VSS is scored out of a total of 13 with a higher score denoting a more severe scar appearance.
The difference in change in acne scar appearance as assessed by the participant using the Vancouver Scar Scale (VSS) between GenLabs' Social Skin and placebo | Day 0 to 20
  The difference in change in acne scar appearance as assessed by the participant using the Vancouver Scar Scale (VSS) between GenLabs' Social Skin and placebo from baseline at Day 20. The VSS is scored out of a total of 13 with a higher score denoting a more severe scar appearance.
The difference in change in acne scar appearance as assessed by the participant using the Vancouver Scar Scale (VSS) between GenLabs' Social Skin and placebo | Day 0 to 30
  The difference in change in acne scar appearance as assessed by the participant using the Vancouver Scar Scale (VSS) between GenLabs' Social Skin and placebo from baseline at Day 30. The VSS is scored out of a total of 13 with a higher score denoting a more severe scar appearance.

OTHER OUTCOMES:
Self-reported incidence of post-emergent adverse events (AE) | Day 0 to 30
  Self-reported incidence of post-emergent adverse events (AE)

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada